CLINICAL TRIAL: NCT02850757
Title: Comparative Study Between Modified William's Airway (Fekry Airway ) Versus the U Shaped Guedl's Airway as Assessed Device for Fiberoptic Intubation.
Brief Title: Comparison Between Modified William's Airway and U Shaped Guedl's Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, lecturer of Anasethiology and pain managment, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N-18-2016
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Endotracheal Intubation
Keywords: Modified William's airway; fiberoptic bronchoscope; U shape Guedls airway; oral airways; efficacy and safety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- U shaped Guedl's airway (Experimental)
  Interventions: Device: U shaped Guedl's airway
- Modified William's airway(Fekry airway ) (Experimental)
  Interventions: Device: Modified William's airway

INTERVENTIONS:
Device: U shaped Guedl's airway — To use U shaped Guedl's airway for assisting fiberoptic bronchoscope during endotracheal intubation
  Arms: U shaped Guedl's airway
Device: Modified William's airway — Use Modified William's airway for assisting fiberoptic bronchoscope dduring endo tracheal intubation
  Other Names: Fekry airway
  Arms: Modified William's airway(Fekry airway )

SUMMARY:
This study will compare the efficacy of modified William's airway versus U shaped Guedl's airway in assistant of fiberoptic bronchoscope during endotracheal intubation

DETAILED DESCRIPTION:
Several oropharyngeal airways and supraglotic devices have been invented to facilitate the art of fiber optic intubation. The oropharyngeal airways help during fiber optic intubation through raising the soft palate and the tongue away from the field of bronchoscope .(1)The modification made to the Williams airway (Fekry's airway) is that the roof of the proximal cylindrical tunnel was removed and opened from its concave part to allow one step insertion of the tube. There is no need for removal of the tube connector or the airway after tube insertion.(3)We invented a new modification in Guedel's airway (The U-shaped Guedel's airway) which is made by making an inverted Y shape cut in the roof of the airway keeping only the proximal Y wings and removing the distal part of the roof.This study will be conducted at Kasr AL-Ainy Hospital Faculty of Medicine Cairo university Egypt , after approval of the ethical committee and taking written informed consents from the patients . Patients presents to the hospital for elective surgery under general anasethia will be randomly divided into 2 groups : Group W (Gw)(n=25 ) the fiber optic intubation will be assisting by modified Williams airway and Group U (Gu)(n=25) the fiber optic intubation will be assisting by U shaped Guedels airway .

In the preparation room 20 guage cannula will be inserted in a peripheral vein . 0,02 mg\ Kg midazolam and 0,01 mg\Kg atropine will be given in the operating room Standard monitors ( ECG, noninvasive Blood pressure and pulse oximetry) will be established to the patient .After 3 minutes preoxygenation with 100% O2 induction was conducted using 1µg\Kg fentanyl,2mg\Kg propofol and 0.05 mg\Kg atracurium. After loss of consciousness the selected airway according to group randomization was inserted into the mouth (size selection and technique of insertion was done according to manufacturer structures . The patient will be ventilated by facemask and bag with 100% oxygen and 1-2% isoflourane. Complete neuromuscular block was confirmed using nerve stimulator (train of four zero).the fiber optic bronchoscope inserted through the airway (modified Williams, U Shaped Guedels airway ) according to the patient group . The time of fiber optic bronchoscope insertion will be recorded in seconds (defined as the time elapsing from the entry of fiber optic bronchoscope through the airway till touching the vocal cords by the tip of bronchoscope) . The investigator will assesse the bronchoscopic view just after the end of the airway . after recording the time of fiberopticbronchoscope insertion the endotracheal tube was slided through vocal cords into the trachea reaching the carina . the patient will be ventilated through the endotracheal tube using intermittent positive pressure ventilation (IPPV) . Endotracheal intubation will be confirmed by chest expansion ,bilateral equal air entry using stethoscope and the appearance 6 successive capnographic waves. Time of intubation will be recorded from stop mask-bag ventilation till reventilate the patient using the endotrachealtube and reading of capnogram. ( the attempt will be cancelled and bag-mask ventilation started if SPO2 reach 93%. )

ELIGIBILITY:
Inclusion Criteria:

* Patient aged above 18 years old.
* Patient that has ASA I,II .
* Patient with Ganzouri airway score less than 4.

Exclusion Criteria:

* Patient aged below 18 years old.
* Patient that has ASA III ,IV.
* Patients at risk of aspiration of gastric content.
* Patient with Ganzouri airway score equal or more than 4.
* Patient that has any anatomical abnormality that invalidate Ganzouri airway score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Time of endotracheal intubation | within 15 minutes from induction of general anesthesia

SECONDARY OUTCOMES:
Time of fiberopticc bronchscpe reach the vocal cords | within 15 minutes from induction of general anesthesia
Bronchoscopic view grade | within 15 minutes from induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Maha My youssef, consultant, Principal Investigator — Kasr alaini hospital,faculty of medicine,cairo university

IPD SHARING:
Plan to Share IPD: No